CLINICAL TRIAL: NCT04556409
Title: Low Intensity Pulsed Ultrasound Therapy Versus Low Level LASER Therapy in the Treatment of Post Cesarean Anterior Cutaneous Branches of Iliohypogastric Neurotmesis
Brief Title: US vs. LASER on Post Cesarean Anterior Cutaneous Branches of Iliohypogastric Neurotmesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohamed Gamal Abouelyazeed Ali, Principal investigator, South Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Post CS numbness
Record Dates: First submitted 2020-09-09; First posted 2020-09-21 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Neurotmesis
Keywords: iliohypogastric neurotmesis; post cesarean; low level laser; low intensity pulsed ultrasound
MeSH Terms: conditions — Trauma, Nervous System

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- low intensity pulsed ultrasound (Experimental): 20 women were treated by low intensity pulsed ultrasound (5 min, 0.5 w/cm2, 1MHZ with 20% duty cycle, 3 times/ week for 4 weeks plus static abdominal and pelvic floor exercises.
  Interventions: Device: low intensity pulsed ultrasound plus static abdominal and pelvic floor exercises.; Other: static abdominal and pelvic floor exercises only.
- low level laser therapy (Experimental): 20 women were treated by low level laser therapy (Gallium Aluminum Arsenide Laser), 808nm, 4J/cm2, pulsating signal, 60 seconds for each point, 30 Mw/cm2, 3 times/week for 4 weeks plus static abdominal and pelvic floor exercises.
  Interventions: Device: low level LASER plus static abdominal and pelvic floor exercises.; Other: static abdominal and pelvic floor exercises only.
- static abdominal and pelvic floor exercises (Placebo Comparator): 20 women were the control group who received only static abdominal and pelvic floor exercises. , 3 times/week for 4 weeks.
  Interventions: Other: static abdominal and pelvic floor exercises only.

INTERVENTIONS:
Device: low intensity pulsed ultrasound plus static abdominal and pelvic floor exercises. — Ultrasonic irradiation was employed with parameters of current use in clinical practice, including lower potency (0.16 W/cm2), which is more adequate for stimulation of nerve regeneration, according to results obtained in investigations in which the irradiation was applied at the lesion site 32, 33.
  Arms: low intensity pulsed ultrasound
Device: low level LASER plus static abdominal and pelvic floor exercises. — Application of laser irradiation (Ga-As laser) in the site of the anastomosis inhibits the degeneration process, accelerate remyelination, and nerve function recovery 27, 28
  Arms: low level laser therapy
Other: static abdominal and pelvic floor exercises only. — static abdominal and pelvic floor exercises., 3 times/week for 4 weeks.

SUMMARY:
the aim of this study is to compare the effect of low intensity pulsed ultrasound therapy and the effect of low level LASER in the treatment of post cesarean anterior cutaneous branches of iliohypogastric neurotmesis.

DETAILED DESCRIPTION:
Cesarean section is one of the commonly performed surgical procedures in obstetrics and is certainly one of the oldest operations in surgery. One of the most dramatic features of modern obstetrics is the increase in the caesarean section rate. In Egypt, the past decade has witnessed a sharp increase in the prevalence of CS with the most recent Egypt Demographic and Health Survey (EDHS) documenting a CS rate of 52%, which suggests that caesarean delivery might be overused or used for inappropriate indications.

Several CS skin incision and abdominal wall opening techniques have been developed during the years, yet a general consensus on the most appropriate approach, in terms of safety and morbidity has not been yet reached 3.The choice of technique depends largely on the Surgeon's experience and preference and on the maternal-fetal clinical condition .

The Pfannenstiel incision and the Misgav-Ladach method, mainly represented by the modified Joel-Cohen incision, are the most common skin incisions performed . The Pfannenstiel incision is a transverse "smile"-like incision made 2-3 cm above the symphysis pubis at the pubic area border; the Misgav-Ladach method is a straight transverse skin incision which lies about 3 cm below the level of the anterior superior iliac spines (ASIS) . Both techniques involve skin and subcutaneous tissues . Although several studies comparing these two abdominal wall opening techniques have been conducted, differences in terms of acute and chronic post-operative pain have not been always considered .

Acute and chronic pain after CS depends mainly on the type of cutaneous incision and subsequent access into the pelvic cavity, in relation to the abdominal wall's somatic innervation .

Both techniques involve an abdominal area innervated by two principal nerves: ileo-hypogastric and ileo-inguinal. These nerves originate from the lumbar plexus, which is formed by the ventral branches of the first to the fourth lumbar nerves (L1-L4) and by the last thoracic nerve (T12) supplementing with a twig .

The iliohypogastric nerve is formed by the fusion of the first lumbar branch with fibers originating from T12. It arises from the upper part of the lateral border of the psoas major then courses infra-laterally atop the quadratus lumborum to the ilium crest where it pierces the transverse abdominal muscle and emerges approximately 3 cm medial to the ASIS. The proximal end of the iliohypogastric nerve enters the abdominal wall 2.8±1.3 cm medial to and 1.4±1.2 cm inferior to the ASIS. Once in the abdominal wall, it follows a linear path terminating 4±1.3 cm lateral to the midline . As the iliohypogastric passes through the abdominal oblique muscles, it divides into the lateral and anterior cutaneous branches which provide sensory innervation to the gluteal (lateral cutaneous branch) and the hypogastric skin regions (anterior cutaneous branch).

For the treatment of peripheral nerve injury, low energy biostimulation lasers are used, applied in the way of pulsatile (905 nm), continuous (808 nm), or pulsing-constant rays. Laser therapy increases the formation of ATP, and the energy of the ATP hydrolysis can be used by nerve cell to restore normal transmembrane potential, which facilitates the generation of electrical impulses and thereby restoring nerve conduction (bioelectric effect). Application of laser beams improves microcirculation and hence nutrition and regeneration of nerve cells - bio-stimulation effect - and increases the release of endorphins and the concentration of neurotransmitters in the synapses - analgetic effect. Application of laser irradiation (Ga-As laser) in the site of the anastomosis inhibits the degeneration process, accelerate remyelination, and nerve function recovery . In the clinic, low-level laser therapy employs doses from 1 to 4J/cm2, associated with output power between 10 to 90mW, and is widely used in various musculoskeletal lesions, as well as in painful and inflammatory processes .

In a precious study had done by Lowdon and Colleagues 30,they found that continous ultrasound at low intensity (0.5W/cm2, 1MHZ, 1min. day every day for 2-3 weeks) was beneficial for regeneration of tibial nerve of rats following compression lesion while continous ultrasound at high intensity (1W/cm2, 1MHZ, 1min. day every day for 2-3 weeks) was harmful for regeneration of tibial nerve of rats following compression injury.

Continous low intensity ultrasound (CLIU) treatment can accelerate the regeneration and functional recovery of neurotometic injured sciatic nerve at earlier stages after injury, the upgraded expression of NGF induced by continuous low intensity ultrasound may be the primary mechanism of the acceleration effects .

ELIGIBILITY:
Inclusion Criteria:

All females were clinically diagnosed with post caesarean anterior cutaneous branches of iliohypogastric neurotmesis by an Obstetrician.

Their ages were ranged from 18 to 35 years old,

All patients participated after removal of surgical stitches (after 2 weeks of cesarean delivery),

All patients were primiparous,

All patients were non-diabetic and all patients received relaxation training.

BMI < 30

Exclusion Criteria:

Multiparous

BMI > 30

Diabetic patients

Smokers

Patients take vitamin B complex

Any previous incision in hypogastric region

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — post cesarean section
Enrollment: 45 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Iliohypogastric nerve injury and recovery | before beginning in the treatment (before the first session) through assessment session the day before beginning the treatment.
  Ultrasonography was used to assess Iliohypogastric nerve injury (pretreatment) and recovery (post treatment) objectively
Iliohypogastric nerve injury and recovery | After last session (after end of the treatment) through one week from last session.
  Ultrasonography was used to assess Iliohypogastric nerve injury (pretreatment) and recovery (post treatment) objectively

SECONDARY OUTCOMES:
sensory function of ilihypogastric nerve | before beginning in the treatment (before the first session) through assessment session the day before beginning the treatment.
  Erasmus MC version of the Nottingham Sensory Assessment was used to assess sensory function of ilihypogastric nerve (pretreatment and posttreatment)
sensory function of ilihypogastric nerve | After last session (after end of the treatment) through one week from last session.
  Erasmus MC version of the Nottingham Sensory Assessment was used to assess sensory function of ilihypogastric nerve (pretreatment and posttreatment)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed GA Ali, Msc, Principal Investigator — Assistant lecturer; Rehab SA Mamoon, Msc, Study Director — Assistant lecturer
Locations (1):
- Faculty of physical therapy, South Valley University, Qina, Qena Governorate, Egypt